CLINICAL TRIAL: NCT02471131
Title: WATCHMAN LAAC Device Implantation During Hybrid Atrial Fibrillation Ablation
Brief Title: WATCHMAN Implantation During Hybrid Ablation
Acronym: WINNING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL.53510.068.15
Record Dates: First submitted 2015-05-20; First posted 2015-06-15 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: WATCHMAN; Atrial Fibrillation; Hybrid Ablation; Safety; Feasibility; Stroke Prevention
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WATCHMAN Implantation (Experimental)
  Interventions: Device: WATCHMAN Device implantation

INTERVENTIONS:
Device: WATCHMAN Device implantation — The implantation of the device will be done into the left atrial appendage according to the guidelines.

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia with a lifetime risk of developing AF of 1 in 4 people aged over 40. Stroke remains the most feared complication of AF with an increase in risk by 5-fold, and is the leading cause of morbidity and mortality. The left atrial appendage (LAA) is the origin for more than 90% of the emboli in non-valvular AF. The WATCHMAN™ Left Atrial Closure Device (WATCHMAN Device, Boston Scientific) reduces the risk of stroke by closing off the LAA. During hybrid procedures for AF, LAA occlusion with epicardial devices is known to be difficult and not free of risks.It thus will be interesting to study the safety and feasibility of endocardial WATCHMAN Device implantation in a hybrid ablation approach.

ELIGIBILITY:
Inclusion Criteria:

* Documented paroxysmal or (long-standing) persistent non-valvular atrial fibrillation,
* Eligible at least for short-term OAC therapy,
* No other conditions that would require long-term OAC therapy, suggested by current standard medical practice, and thus is eligible to stop OAC if the LAA is sealed,
* Calculated CHA2DS2-VASc score of 1 or more,
* 18 years of age or older, able and willing to provide written informed consent.

Exclusion Criteria:

* Current New York Heart Association Class IV Congestive Heart Failure,
* Current thrombocytopenia (< 100x10E9/L) or anemia (hemoglobin <6.2 mmol/L),
* Active infection or sepsis,
* Resting heart rate > 110 beats per minute,
* Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the last 30 days,
* Recent myocardial infarction (within 3 months),
* Transient case of AF (i.e., secondary to recent cardiac surgery (within 3 months)),
* Planned cardioversion 30 days post implant of the WATCHMAN Device,
* Implanted mechanical valve prosthesis,
* History of obliterated LAA,
* History of heart transplantation,
* Symptomatic carotid disease (i.e., carotid stenosis >50% associated with ipsilateral transient or visual ischemic attack evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke within 6 months),
* Necessity to use long-term OAC,
* Contraindication for use of OAC or dual anti-platelet therapy,
* Contraindication for use of aspirin,
* Pregnancy or planned pregnancy during the course of the investigation,
* Life expectancy less than 2 years,
* Participation in any other clinical study involving an investigational drug or device.

Echocardiographic Exclusion Criteria (as assessed via transthoracic echocardiography (TTE) or TEE) for this study are:

* Left ventricular ejection fraction (LVEF) < 30%,
* Intracardiac thrombus as visualized by TEE within 2 days prior to implant,
* High risk patent foramen ovale,
* Current atrial septal defect and/or previous atrial septal repair or closure device,
* Significant mitral valve stenosis (i.e., MV 4. 5 cm2),
* Existing pericardial effusion of >3 mm,
* Complex atheroma with mobile plaque of the descending aorta and/or aortic arch,
* Cardiac tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Major complications during follow-up, assessed by scoring the number of complications | 6 months
Device success, assessed by transesophageal echocardiogram. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pison, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Vroomen M, Maesen B, Luermans JG, Crijns HJ, Maessen JG, La Meir M, Pison L. Left Atrial Appendage Management with the Watchman Device during Hybrid Ablation of Atrial Fibrillation. J Interv Cardiol. 2019 Jun 26;2019:4525084. doi: 10.1155/2019/4525084. eCollection 2019. PMID 31772531